CLINICAL TRIAL: NCT05499247
Title: A Proof-of-Concept, Safety and Efficacy Study of SkinQ Glow Bright Wonder Mask in Healthy Human Subjects and With Adequate Representation of Varied Skin Types (Normal, Oily, Dry, Combined, and Sensitive Skin)
Brief Title: A Proof-of-Concept, Safety and Efficacy Study of SkinQ Glow Bright Wonder Mask in Healthy Human Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NovoBliss Research Pvt Ltd (Other)
Responsible Party: Principal Investigator, Dr Nayan Patel, Principal Investigator, NovoBliss Research Pvt Ltd
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NB220018-SQ
Record Dates: First submitted 2022-08-03; First posted 2022-08-12 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Healthy Human Volunteers With Visibly Tanned Skin
Keywords: Healthy; Tanned Skin

STUDY DESIGN:
Intervention Model Description: Proof-of-Science, Safety and Efficacy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental)
  Interventions: Other: SkinQ Glow Bright Wonder Mask

INTERVENTIONS:
Other: SkinQ Glow Bright Wonder Mask — Mode of Usage:
  Cleanse and dry face. Apply 1 tsp or 5g of the product. Apply with clean finger or brush to full face. Leave to dry for 15 minutes. Wipe with wet cotton or rinse with cool water.
  Route of Administration: Topical

SUMMARY:
This is an open-label, single-arm, single-centre, proof-of-concept, safety and efficacy, clinical study of SkinQ Glow Bright Wonder Mask in Healthy Human Subjects and adequate representation of varied skin types [Normal, Oily, Dry, Combined and Sensitive skin].

The rationale of the study is to evaluate whether the product SkinQ Glow Bright Wonder Mask is providing an instant skin tanning reduction in 15 mins, smoother, softer and glows skin, and even/brighter complexion in 15 mins, instant improvement in skin brightness and not just a marketing gimmick. It is also to assess the efficacy of the product in its performance for the following parameters:

* Tan reduction
* Close pores
* Makes skin bright and radiant.
* Removes tan marks
* Fades dark spots of pimple and acne
* Gives a glowing look
* The texture of the product, experience, acceptability

DETAILED DESCRIPTION:
The potential subjects will be screened as per the inclusion & exclusion criteria only after obtaining written informed consent from the subjects. This is a single-day, single-visit study.

Subjects will be pre-screened by the screening department of NovoBliss Research. Subjects will be called on the telephone by the recruiting department prior to the enrolment visit. They will be asked a series of questions that are provided on the Screener Form (an example template is provided in Appendix III). This form will be saved electronically, and if subjects are eligible for the study as determined by the responses given on the Screener Form, subjects may be asked to participate in the enrolment visit. Subjects will be told during screening (prior to enrolment) not to wear any facial make-up on the study visit day. It is also recommended that the subjects are told to bring a hair tie to pull their hair back if desired during the study.

Assessment of efficacy parameters before application, after product removal at 5 mins, 15mins will be done on day 1 of the study as listed below.

* Skin ColorimeterCL- 400 (Courage Khazaka Instrument): (International Commission on Illumination) CIE L-, a-, b- value, ITA (Individual Topology Angle] - instant change in skin colour, tone
* Visioscan®VC20plus - SELS (Surface Evaluation of the Living Skin), Pores - Skin Surface Assessment: Roughness, smoothness, texture
* 3D Imaging Pictures
* Sensorial Evaluation-- Subjective evaluation of skin brightness, and skin tanning: on a four-point scale (absent, mild, moderate, or severe)
* Digital Photographs: Before Application and after product removal.
* Local irritation (erythema, scaling, itching, and burning): using a four-point scale (absent, mild, moderate, severe)
* Skin pigmentation scoring
* Subjects Response Index [Consumer Perception about Product] Before Application and After product removal

  * Product acceptance related to physical properties (consistency, colour, fragrance) on five-point scale
  * Product acceptance related to cosmetic properties (spreadability, permeability and fixation) on five-point scale
  * Subjects Satisfaction with cosmetic properties

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 to 55 years (both inclusive) old at the time of consent.
2. Sex: Healthy adult males and non-pregnant/non-lactating females.
3. Subject with normal Fitzpatrick skin type III to VI (Human skin colour determination scale).
4. Females of childbearing potential must have a self-reported negative urine pregnancy test.
5. Subjects are generally in good general health as determined from recent medical history.
6. Subjects with visibly tanned skin determine by a dermatologist or dermatologist trained evaluator.
7. The subject does not have any previous history of adverse skin conditions and is not under any medication likely to interfere with the results.
8. The subjects who have not done any facial treatment, or any herbal facial, tanning removal for more than 30 days and who regularly use tanning removal products.
9. The subject is willing and able to follow the study directions, and participate in the study.
10. The subject must be able to understand and provide written informed consent to participate in the study.

Exclusion Criteria:

1. Subject with known allergy or sensitization to product ingredients such as niacinamide, glycolic acid, Liquorice, vitamin c, mulberries, purple brazilian clay or any other ingredients.
2. The subject had a facial or chemical peeling or derma abrasion | roller etc. in the last 4 weeks.
3. The subject has skin irritation, open wounds, cuts, abrasions, irritation symptoms or any dermatological condition on the face that can interfere with the reading.
4. Be wearing any facial makeup, including false eyelashes, on the day of the study visit.
5. Be using any skin lightening | brightening or tanning removal product within 15 days and on the day of the study visit.
6. Medication which may affect skin response and/or past medical history.
7. The subject has a history of diabetes
8. The subject has a history of mastectomy for cancer involving removal of lymph nodes within the past year, or treatment of any type of cancer within the last 6 months.
9. The subject suffering from any active clinically significant skin diseases which may contraindicate.
10. The subject has a history of any skin diseases including eczema, atopic dermatitis etc.
11. Subject with self-reported immunological disorders such as HIV positive, AIDS and/or systemic lupus erythematosus.
12. Have taken antihistamines (including those in cold tablets, OTC (over-the-counter) allergy medications, decongestants and inhalants) or analgesics (including aspirin or other over-the-counter analgesics) on the days of the study.
13. An individual who has a medical condition or is taking or has taken a medication which, in the Investigator's judgment, makes the subject ineligible or places the subject at undue risk.
14. Participation in other clinical studies simultaneously.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2022-08-29 (Actual); Primary Completion 2022-09-06 (Actual); Study Completion 2022-09-14 (Actual)

PRIMARY OUTCOMES:
To assess the instant change in skin colour, and tone | On Day 01 before application and after product removal at 5 mins and 15 mins
  To assess the instant change in skin colour, and tone with a single application of the test product using Skin ColorimeterCL-400 by measuring CIE (International Commission on Illumination) L-, a-, b- value, ITA (Individual Topology Angle)
Surface evaluation of the living skin SELS® (Surface Evaluation of the Living Skin) | On Day 01 before application and after product removal at 5 mins and 15 mins
  To assess the instant change in skin surface i.e. smoothness, roughness, scaliness, wrinkles based on the grey levels of the image in a single application using Visioscan®VC20plus
To assess the instant change in skin pores | from the baseline on Day 01 before application and after product removal at 5 mins and 15 mins
  To assess the instant change in skin pores in a single application using Visioscan®VC20plus

SECONDARY OUTCOMES:
Instant change in skin brightness, skin tanning | on Day 01 before application and after product removal at 15 mins
  To assess the effect of the test product in terms of instant change in skin brightness, skin tanning in a single application by dermatologist trained evaluator or dermatologist
Local Irritation (erythema, scaling, itching, and burning) | On Day 01 before application and after product removal at 15 mins
  To assess the effect of the test product in terms of local irritation (erythema, scaling, itching, and burning) in a single application by dermatologist trained evaluator or dermatologist
Skin Pigmentation | On Day 01 before application and after product removal at 15 mins
  To assess instant change in skin pigmentation in a single application by dermatologist trained evaluator or dermatologist
Sensorial Evaluations | Before product application and after 15 mins of post product removal
  Subjective perception questionnaires on the sensorial evaluations of test product will be asked by study staff after the removal of product on physical properties of the product i.e. consistency, colour, fragrance; product cosmetics properties i.e. spreadability, permeability, fixation, and product usage on skin tan reduction, skin brightening, radiance, fading dark spots, glowing skin, smoothness, roughness, scaliness, feel about burning, redness, itching, tingling upon product application

OTHER OUTCOMES:
Treatment Emergent adverse events | On Day 01 after product application and removal
  Safety will be determined by treatment-emergent adverse events such as unbearable irritation, redness, tingling, dryness of skin, and burning sensation assessed by the Dermatologist or Study Physician

CONTACTS AND LOCATIONS:
Overall Officials: Dr Nayan K Patel, MBBS, Principal Investigator — Medical Director
Locations (1):
- NovoBliss Research Pvt Ltd, Gandhinagar, Gujarat, India

IPD SHARING:
Plan to Share IPD: No